CLINICAL TRIAL: NCT03919994
Title: OASIS: Observational Study of LAIs In Schizophrenia
Brief Title: Observational Study of Long Acting Injectable Medications (LAIs) in Schizophrenia (OASIS)
Status: Completed | Type: Observational
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALKS 9072-A403N
Record Dates: First submitted 2019-04-01; First posted 2019-04-18 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
Keywords: Alkermes; Schizophrenia; ARISTADA; Abilify Maintena; Invega Sustenna; Risperdal Consta; Cohort Study; Observational; Phase 4
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (4):
- ABILIFY MAINTENA®: Subjects newly initiated
- ARISTADA®: Subjects newly initiated
- INVEGA SUSTENNA®: Subjects newly initiated
- RISPERDAL CONSTA®: Subjects newly initiated

SUMMARY:
The objectives of this study are to describe characteristics, treatment patterns, and outcomes of patients with schizophrenia newly initiated on 1 of 4 FDA-approved atypical Long Acting Injectable (LAI) antipsychotics (ABILIFY MAINTENA®, ARISTADA®, INVEGA SUSTENNA® or RISPERDAL CONSTA®)

DETAILED DESCRIPTION:
This is a non-interventional, prospective, multi-center observational cohort study. Patients at behavioral health clinics will be enrolled and evaluated by health care professionals (e.g., psychiatrists) according to the standard of care. All patients will be followed for approximately 12 months from their enrollment visit.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to speak, read and understand English
* Diagnosis of schizophrenia as defined by the treating clinician
* Newly initiating treatment with 1 of 4 atypical Long Acting Injectables (LAIs): Abilify Maintena, Aristada, Invega Sustenna, or Risperdal Consta)
* Additional criteria may apply

Exclusion Criteria:

* Currently participating or planning to participate in an interventional clinical study, or has completed participation in an interventional clinical study within 30 days before enrollment
* In the opinion of the investigator, is currently an imminent danger to himself/herself. [Note: A prior history of suicidal ideation or suicidal attempt is not exclusionary.]
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia who are newly initiating LAI treatment
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Schizophrenia disease history | Baseline
  Including time (years) since diagnosis as assessed from clinical history
Number of comorbid conditions at baseline | Baseline
  Assessed from clinical history
Changes in comorbid conditions | Up to 12 months
  The percent of patients experiencing each comorbid condition will be assessed at follow-up visits
Number of LAI injections | Up to 12 months
  Average number of injections during treatment period
Number of patients switching or discontinuing LAI treatment | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (52):
- United States (52):
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Costa Mesa, California
  - Alkermes Investigational Site, El Cajon, California
  - Alkermes Investigational Site, Granada Hills, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Panorama City, California
  - Alkermes Investigational Site, San Bernardino, California
  - Alkermes Investigational Site, Dayville, Connecticut
  - Alkermes Investigational Site, Hialeah, Florida
  - Alkermes Investigational Site, Lauderdale Lakes, Florida
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigational Site, Miami Gardens, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, Panama City, Florida
  - Alkermes Investigational Site, Tallahassee, Florida
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Lawrenceville, Georgia
  - Alkermes Investigational Site, Honolulu, Hawaii
  - Alkermes Investigational Site, Schaumburg, Illinois
  - Alkermes Investigational Site, Springfield, Illinois
  - Alkermes Investigational Site, Indianapolis, Indiana
  - Alkermes Investigational Site, Bel Air, Maryland
  - Alkermes Investigational Site, Boston, Massachusetts
  - Alkermes Investigational Site, Grand Rapids, Michigan
  - Alkermes Investigational Site, Kalamazoo, Michigan
  - Alkermes Investigational Site, Kansas City, Missouri
  - Alkermes Investigational Site, Raymore, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Lincoln, Nebraska
  - Alkermes Investigational Site, Manchester, New Hampshire
  - Alkermes Investigational Site, Buffalo, New York
  - Alkermes Investigational Site, Glen Oaks, New York
  - Alkermes Investigational Site, Jamaica, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Poughkeepsie, New York
  - Alkermes Investigational Site, Beachwood, Ohio
  - Alkermes Investigational Site, Fairlawn, Ohio
  - Alkermes Investigational Site, Westlake, Ohio
  - Alkermes Investigational Site, Wooster, Ohio
  - Alkermes Investigational Site, Durant, Oklahoma
  - Alkermes Investigational Site, Tulsa, Oklahoma
  - Alkermes Investigational Site, Eugene, Oregon
  - Alkermes Investigational Site, Wyomissing, Pennsylvania
  - Alkermes Investigational Site, Sioux Falls, South Dakota
  - Alkermes Investigational Site, Franklin, Tennessee
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Fort Worth, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Richmond, Texas
  - Alkermes Investigational Site, San Antonio, Texas
  - Alkermes Investigational Site, Wichita Falls, Texas
  - Alkermes Investigational Site, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haider B, O'Sullivan AK, Bessonova L, Keane E, Achtyes E, Harvey PD, Kane JM, Saklad SR, Trotter JP, Claxton A, Polak T, McGrory J, Noori W, Sikora Kessler A, Yarlas A, Velligan D. Changes in Clinical Management of Patients with Schizophrenia Treated with Long-Acting Injectable Antipsychotics (LAIs), Including Telepsychiatry Use, During the COVID-19 Pandemic. Neuropsychiatr Dis Treat. 2023 Mar 17;19:623-634. doi: 10.2147/NDT.S394220. eCollection 2023. PMID 36959874